CLINICAL TRIAL: NCT02127242
Title: The Study of Laparoscope Combined Ureteroscopic Air-pressure Ballistic Lithotripsy to Treat Patients With Hepatolithiasis
Brief Title: Laparoscope Combined Ureteroscopic Air-pressure Ballistic Lithotripsy to Treat Patients With Hepatolithiasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fanyingfang2
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Cholelithiasis
Keywords: hepatolithiasis; ureteroscope; air-pressure ballistic lithotripsy; hepatectomy
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- air-pressure ballistic lithotripsy (Experimental): In case of large, hard or impacted stones ureteroscopic air-pressure ballistic lithotripter is used for fragmentation. The probe of the lithotripter target towards the stone and then fragmented.
  Interventions: Procedure: ureteroscopic air-pressure ballistic lithotripsy
- hepatectomy group (No Intervention): Hepatic resection using an open approach is performed for all segments affected by biliary stenosis and the affected bile duct drainage area.Hepaticojejunostomy is performed in patients with common bile duct stenosis and in those considered to be at high risk for recurrence.

INTERVENTIONS:
Procedure: ureteroscopic air-pressure ballistic lithotripsy — In case of large, hard or impacted stones ureteroscopic air-pressure ballistic lithotripter is used for fragmentation. The probe of the lithotripter target towards the stone and then fragmented.
  Other Names: UAPBL
  Arms: air-pressure ballistic lithotripsy

SUMMARY:
Objective:the purpose of this study is to investigate the efficacy,feasibility,reliability,and safety of laparoscope combined air-pressure ballistic lithotripsy in the treatment of patients with bile duct stones.

Methods:We are going to select 60 patients diagnosed with hepatolithiasis who carry on the treatment in our hospital from April 2014 to April 2015.According to the unified inclusion and exclusion criteria,the patients are divided into the experimental group and the control group.The experimental group use the treatment of laparoscope combine with air-pressure ballistic lithotripsy to treat hepatolithiasis,while the control group treat the patients with hepatolithiasis with the method of lobectomy and segmental resection of liver.Contrastive analyzed two group of patients' clinical care effects.

Research hypothesis:according to compare two groups' duration of surgery,blood loss,postoperative complication rate,hospital stay,the stone clearance rate,,the residual stone rate,reoperation rate etc.We suppose that the clinical results of the experimental group are superior to the control group,difference is statistically significant(P<0.05).So we can draw the conclusion that the method of laparoscope combined air-pressure ballistic lithotripsy is useful in treatment of patients with hepatolithiasis.

DETAILED DESCRIPTION:
To select 60 patients diagnosed with hepatolithiasis who carry on the treatment in our hospital from April 2014 to April 2015.According to the unified inclusion and exclusion criteria,the patients are divided into the experimental group and the control group.The experimental group use the treatment of laparoscope combine with air-pressure ballistic lithotripsy to treat hepatolithiasis,while the control group treat the patients with hepatolithiasis with the method of lobectomy and segmental resection of liver.

The experimental group performed under the situation of tracheal intubation general,placing the ureteroscope into common bile duct and exploring the bile duct after laparoscopic cholecystectomy and choledochotomy.Associated with air-pressure ballistic lithotripsy once discover bile duct stones and retrieve the rubble by flowing it out.To stone's diameter lower than 5 mm,use lithotomy forceps pull it out.Examining the bottom of common bile duct,ensuring that it will not obstructed.Last,placing the T-tube continuous drainage the residual stones.The control group using the way of hepatectomy.Choosing suitable surgical options according to the stones' location and associating with choledochoenterostomy if needed.

Contrastive analyse two groups' clinical indicators,such as operation time,blood loss during the surgery,hospital stay,the stone clearance rate,the residual stone rate,the incidence of postoperative complications and so on.

.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatolithiasis;
* Patients with hepatolithiasis and extrahepatic bile duct stones or gallbladder stones;
* Patients with hepatolithiasis and acute cholangitis whose inflammation subside more than one month by conservative therapy.
* Regularly visiting our hospital;
* Willing to comply with all study procedures and provided signed and dated informed consent.

Exclusion Criteria:

* Simply gallbladder stones;
* Hepatolithiasis with carol's disease;
* Hepatolithiasis with bile duct carcinoma;
* patients with the clinical performances of severe cholangitis;
* patients with biliary stricture obviously;
* patients with heart,lungs,hepatic or renal dysfunction.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-03 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
residual stone rate | 2 weeks
the stone clearance rate | 2 weeks

SECONDARY OUTCOMES:
the incidence of postoperative complications | one month

OTHER OUTCOMES:
reoperation rate | one month

CONTACTS AND LOCATIONS:
Overall Officials: Fan y fang, Prof., Principal Investigator — Department of Hepatobiliary Surgery(I),Zhujiang Hospital
Locations (1):
- Department of Hepatobiliary (I),Zhujiang Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Farooq Qadri SJ, Khan M, Khan N. Use of pneumatic lithotripsy for managing difficult CBD calculi. Int J Surg. 2011;9(1):59-62. doi: 10.1016/j.ijsu.2010.08.009. Epub 2010 Sep 16. PMID 20849989